CLINICAL TRIAL: NCT00947765
Title: Phase 2/Phase 3 of the Randomized Control Trial to Evaluate the Efficacy of Autologous Blood Injection Versus Local Corticosteroid Injection for Treatment of Lateral Epicondylitis.
Brief Title: A Randomized Control Trial to Evaluate the Efficacy of Autologous Blood Injection Versus Local Corticosteroid Injection for Treatment of Lateral Epicondylitis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Dojode, Chetan M., MBBS, MS (Individual)
Responsible Party: Dr. Chetan Muralidhara Rao Dojode, MBBS,MS(Ortho), Dr. Chetan Muralidhara Rao Dojode. Resident in Orthopaedics and Traumatology.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Lateralepicondylitis- ChetanMD
Record Dates: First submitted 2009-07-27; First posted 2009-07-28 (Estimated); Results first posted 2010-07-23 (Estimated); Last update posted 2010-07-28 (Estimated); Status verified 2009-10

CONDITIONS: Tennis Elbow; Epicondylitis, Lateral Humeral
Keywords: Tennis Elbow; Epicondylitis, Lateral Humeral
MeSH Terms: conditions — Tennis Elbow

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Autologous blood injection group (Experimental): This is the study group in whom autologous blood injection was injected at lateral epicondylitis site.
  Interventions: Biological: Autologous blood injection
- Local corticosteroid injection group (Active Comparator): This is the control group in whom the commonly used treatment modality-local corticosteroid injection was given at lateral epicondyle site.
  Interventions: Drug: Local corticosteroid injection

INTERVENTIONS:
Biological: Autologous blood injection — Patients were infiltrated with injection of 2 ml autologous blood drawn from contra lateral upper limb vein mixed with 1 ml 0.5% bupivacaine, at the lateral epicondyle according to the standard technique.
  Other Names: autologous blood drawn from peripheral vein.
  Arms: Autologous blood injection group
Drug: Local corticosteroid injection — Patients were infiltrated with 2 milliliters of local corticosteroid (Methyl prednisolone acetate 80mg) mixed with 1 milliliters 0.5% Bupivacaine, at the lateral epicondyle according to the standard technique
  Other Names: Methyl prednisolone acetate 80mg
  Arms: Local corticosteroid injection group

SUMMARY:
Lateral epicondylitis, is a common problem encountered in the orthopaedic practice. Histopathological reports have shown that lateral epicondylitis is not an inflammatory process but a degenerative condition termed 'tendinosis'. Beneficial effects of local corticosteroid infiltration have sound lack of scientific rationale, since surgical specimens show lack of any inflammatory process. Recently an injection of "autologous blood injection" has been reported to be effective for both intermediate and long term outcomes. It is hypothesized that blood contains platelet derived growth factor induce fibroblastic mitosis and chemotactic polypeptides such as transforming growth factor cause fibroblasts to migrate and specialize and have been found to induce healing cascade. The objective of the study is to evaluate the efficacy of autologous blood injection versus local corticosteroid injection in the management of lateral epicondylitis.

DETAILED DESCRIPTION:
Much controversy has been there over the pathophysiology and there is not enough scientific evidence to favour any particular type of treatment for acute lateral epicondylitis. Currently degeneration of the origin of the extensor carpi radialis brevis (ECRB), repeated micro trauma and incomplete healing response has been accepted as the cause of lateral epicondylitis by most of the researchers.

Histopathological reports have shown that lateral epicondylitis is not an inflammatory process but a degenerative condition termed 'tendinosis'. There are numerous treatment modalities for lateral epicondylitis both conservative and operative. Most conservative modalities such as local corticosteroid injection have focused on suppressing inflammatory process that does not actually exist. A recent review article concluded that for short term outcomes (6 weeks), statistically significant and clinically relevant differences were found on pain and global improvement with corticosteroid injection compared to placebo, local anaesthetic, or other conservative treatments. For intermediate (6 weeks to 6 months) and long term outcomes (more than 6 months), no statistically significant or clinically relevant results in favour of corticosteroid injections were found. So it is not possible to draw a firm conclusion on the effectiveness of corticosteroid injection.

Recently an injection of autologous blood has been reported to be effective for both intermediate and long term outcomes for the treatment of lateral epicondylitis. There was a significant decrease in pain. It is hypothesized that mitogens such as platelet derived growth factor induce fibroblastic mitosis and chemotactic polypeptides such as transforming growth factor cause fibroblasts to migrate and specialize and have been found to cause angiogenesis. A specific humoral mediator may promote the healing cascade in the treatment of tendinosis as well. These growth factors trigger stem cell recruitment, increase local vascularity and directly stimulate the production of collagen by tendon sheath fibroblasts.

Autologous blood was selected as the medium for injection because (1) its application is minimally traumatic, (2) it has a reduced risk for immune-mediated rejection, devoid of potential complications such as hypoglycemia, skin atrophy, tendon tears associated with corticosteroid injection (3) it is simple to acquire and prepare, easy to carry out as outpatient procedure and (4) it is inexpensive.

There are very few studies done to evaluate injection of autologous blood for lateral epicondylitis as treatment modality. Hence it is evaluated by comparing with the corticosteroid injection which is a commonly practiced conservative treatment modality.

ELIGIBILITY:
Inclusion Criteria:

1. Cases of lateral epicondylitis.
2. Men and women above fifteen years of age.

Exclusion Criteria:

1. Patients receiving steroid injections within three months before blood injection.
2. A history of substantial trauma.
3. Previously treated by surgery for lateral epicondylitis.
4. Other causes of elbow pain such as osteochondritis dessecans of capitellum, lateral compartment arthrosis, varus instability, radial head arthritis, posterior interosseous nerve syndrome, cervical disc syndrome, synovitis of radiohumeral joint, cervical radiculopathy, fibromyalgia, osteoarthritis of elbow, carpel tunnel syndrome.

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-01; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Vijay kumar G Murakibhavi, MS(Ortho), Study Chair — Professor of Orthopaedics. Jawaharlal Nehru Medical College. Belgaum. Karnataka. India.; Dr. Chetan M Dojode, MBBS,MS(Ortho), Study Chair — Senior Resident (Dept. of Orthopaedic and Traumatology)
Locations (1):
- Jawaharlal Nehru Medical College. KLES Dr.Prabhakar Kore Hospital and Medical Research Center., Belagavi, Karnataka, India

REFERENCES:
- [Result] Edwards SG, Calandruccio JH. Autologous blood injections for refractory lateral epicondylitis. J Hand Surg Am. 2003 Mar;28(2):272-8. doi: 10.1053/jhsu.2003.50041. PMID 12671860
- See also: Sonographic-guided blood injection has been reported to improve clinical outcome. It can also be used to monitor the changes to the common extensor origin — http://www.ncbi.nlm.nih.gov/pubmed/16552606
- See also: Autologous preparations rich in growth factors promote proliferation and induce VEGF and HGF production by human tendon cells in culture. — http://www.ncbi.nlm.nih.gov/pubmed/15779147

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were selected by interview and clinical examination and Consent was taken.
  Location: Out patient department of KLES Dr. Prabhakar Kore Hospital & MRC, Belgaum.
  Period: January 1st, 2007-December 31st, 2007. No blinding procedure was followed. Randomization: participants were assigned into two groups according to randomization table.
Period: Overall Study
Arm/Group | Autologous Blood Injection Group | Local Corticosteroid Injection Group
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Autologous Blood Injection Group | Local Corticosteroid Injection Group | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1
  Between 18 and 65 years | 28 | 29 | 57
  >=65 years | 2 | 0 | 2
Age Continuous [Mean (Standard Deviation); unit: years] | 42.9 (12.7721) | 42.3 (9.51) | 42.6 (11.1678)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 18 | 35
  Male | 13 | 12 | 25
Region of Enrollment [Number; unit: participants]
  India | 30 | 30 | 60
Laterality of limb involved [Number; unit: participants] — Participants with Right limb involved / Participants with Left limb involved
  participants
    Participants with Right limb involved | 23 | 23 | 46
    Participants with Left limb involved | 7 | 7 | 14
Participants with Dominant and Non-Dominent limb involvement [Number; unit: participants] — Participants with Dominant limb involved / Participants with Non-Dominent limb involved
  participants
    Participants with Dominent limb involved | 25 | 26 | 51
    Participants with Non-Dominant limb involved | 5 | 4 | 9
Pain: Nirschl Staging (0 to 7) [Mean (Standard Deviation); unit: Units on a scale] — NIRSCHL STAGING:
  phase1: mild pain with exercise; resolves within 24 hours phase2: pain after exercise; exceeds 48 hours phase3: pain with exercise; does not alter activity phase4: pain with exercise; alters activity phase5: pain with heavy activities of daily living phase6: pain with light activities of daily living; intermittent pain at rest phase7: constant pain at rest; disrupts sleeps No pain______1 ______ 2______ 3_______4______ 5______ 6 _____ 7 worst pain
  Units on a scale | 5.4 (1.1325) | 5.23 (0.9714) | 5.315 (1.049)
Pain: Visual Analogue Scale (0 to 10) [Mean (Standard Deviation); unit: Units on a scale] — PAIN SCORE; VISUAL ANALOGUE SCALE:
  Pain of the participants will be assessed by most widely used and accepted "visual analogue scale". It consists of a 10 centimeter line marked at one end with "no pain" and at other end with "worst pain ever". Participant is asked to indicate where on the line he or she rates the pain on the day of presentation, 1, 4, 12weeks and 6 month of follow-ups. Numerical valve is then given to it simply by measuring length between "no pain" to patients mark.
  No pain____1___2___3___4___5___6___7___8___9___10 worst pain ever.
  Units on a scale | 7.7 (1.3429) | 7.533 (1.2794) | 7.616 (1.303)

OUTCOME MEASURES:

1. Primary Outcome: Pain (at 1 Week): Visual Analogue Scale(0 to 10)
Description: VISUAL ANALOGUE SCALE:
  Pain of the participants will be assessed by most widely used and accepted "visual analogue scale". It consists of a 10 centimeter line marked at one end with "no pain" and at other end with "worst pain ever". Participant is asked to indicate where on the line he or she rates the pain on the day of presentation, 1, 4, 12weeks and 6 month of follow-ups. Numerical valve is then given to it simply by measuring length between "no pain" to patients mark.
  No pain____1___2___3___4___5___6___7___8___9___10 worst pain ever.
Time Frame: 1 week
Population: Participants were clinically examined for the treatment response i.e., decrease in pain.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Autologous Blood Injection Group | Local Corticosteroid Injection Group
Number analyzed (Participants) | 30 | 30
Units on a scale | 7.166 (1.9312) | 4.5 (1.8708)
Statistical Analysis 1: Comparison: Autologous Blood Injection Group vs Local Corticosteroid Injection Group; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Pain(at 1 Week): Nirschl Staging (0 to 7)
Description: NIRSCHL STAGING:
  phase1: mild pain with exercise; resolves within 24 hours phase2: pain after exercise; exceeds 48 hours phase3: pain with exercise; does not alter activity phase4: pain with exercise; alters activity phase5: pain with heavy activities of daily living phase6: pain with light activities of daily living; intermittent pain at rest phase7: constant pain at rest; disrupts sleeps
  No pain______1 ______ 2______ 3_______4______ 5______ 6 _____ 7 worst pain
Time Frame: 1 week
Population: Participants were clinically examined for the treatment response i.e., decrease in pain.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Autologous Blood Injection Group | Local Corticosteroid Injection Group
Number analyzed (Participants) | 30 | 30
Units on a scale | 5.1 (1.4703) | 3.06 (1.3629)
Statistical Analysis 1: Comparison: Autologous Blood Injection Group vs Local Corticosteroid Injection Group; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney)

3. Primary Outcome: Pain(at 4 Weeks): Visual Analogue Scale
Description: VISUAL ANALOGUE SCALE:
  Pain of the participants will be assessed by most widely used and accepted "visual analogue scale". It consists of a 10 centimeter line marked at one end with "no pain" and at other end with "worst pain ever". Participant is asked to indicate where on the line he or she rates the pain on the day of presentation, 1, 4, 12weeks and 6 month of follow-ups. Numerical valve is then given to it simply by measuring length between "no pain" to patients mark.
  No pain____1 ___ 2 ___ 3 ___ 4 ___ 5 ___ 6 ___ 7 ___ 8 ___ 9 ___ 10 worst pain ever.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Autologous Blood Injection Group | Local Corticosteroid Injection Group
Number analyzed (Participants) | 30 | 30
Units on a scale | 3.2 (2.369) | 1.533 (2.315)
Statistical Analysis 1: Comparison: Autologous Blood Injection Group vs Local Corticosteroid Injection Group; Test type: Superiority or Other; p = 0.0022, Wilcoxon (Mann-Whitney)

4. Primary Outcome: Pain(at 4 Weeks): Nirschl Staging
Description: as for outcome 2
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Autologous Blood Injection Group | Local Corticosteroid Injection Group
Number analyzed (Participants) | 30 | 30
Units on a scale | 2.2 (1.6484) | 1.03 (1.5862)
Statistical Analysis 1: Comparison: Autologous Blood Injection Group vs Local Corticosteroid Injection Group; Test type: Superiority or Other; p = 0.003, Wilcoxon (Mann-Whitney)

5. Primary Outcome: Pain(at 12 Weeks): Visual Analogue Scale
Description: as for outcome 3
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Autologous Blood Injection Group | Local Corticosteroid Injection Group
Number analyzed (Participants) | 30 | 30
Units on a scale | 0.6 (1.9046) | 1.5 (1.8147)
Statistical Analysis 1: Comparison: Autologous Blood Injection Group vs Local Corticosteroid Injection Group; Test type: Superiority or Other; p = 0.0127, Wilcoxon (Mann-Whitney)

6. Primary Outcome: Pain(at 12 Weeks): Nirschl Staging
Description: as for outcome 2
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Autologous Blood Injection Group | Local Corticosteroid Injection Group
Number analyzed (Participants) | 30 | 30
Units on a scale | 0.433 (1.278) | 1.03 (1.3257)
Statistical Analysis 1: Comparison: Autologous Blood Injection Group vs Local Corticosteroid Injection Group; Test type: Superiority or Other; p = 0.0184, Wilcoxon (Mann-Whitney)

7. Primary Outcome: Pain(at 6 Months): Visual Analogue Scale
Description: as for outcome 3
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Autologous Blood Injection Group | Local Corticosteroid Injection Group
Number analyzed (Participants) | 30 | 30
Units on a scale | 0.533 (1.907) | 1.833 (2.0356)
Statistical Analysis 1: Comparison: Autologous Blood Injection Group vs Local Corticosteroid Injection Group; Test type: Superiority or Other; p = 0.0058, Wilcoxon (Mann-Whitney)

8. Primary Outcome: Pain(at 6 Months): Nirschl Staging
Description: as for outcome 2
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Autologous Blood Injection Group | Local Corticosteroid Injection Group
Number analyzed (Participants) | 30 | 30
Units on a scale | 0.366 (1.2726) | 1.233 (1.4308)
Statistical Analysis 1: Comparison: Autologous Blood Injection Group vs Local Corticosteroid Injection Group; Test type: Superiority or Other; p = 0.0064, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Follow up was done up to 6 months.
Arm/Group | Autologous Blood Injection Group | Local Corticosteroid Injection Group
Serious Adverse Events (participants affected / at risk) | 0/30 | 2/30
Other Adverse Events (participants affected / at risk) | 0/0 | 0/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Autologous Blood Injection Group (N=30) | Local Corticosteroid Injection Group (N=30)
Elbow stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0)
Infection (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0)
Injury to cutanous nerve (Nervous system disorders) | 0 (0) | 0 (0)
Local skin atrophy (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Autologous Blood Injection Group (N=0) | Local Corticosteroid Injection Group (N=30)
Systemic affects of Corticosteroid injection (Endocrine disorders) | 0 (0) | 0 (0) — This adverse event is assesed only in Local corticosteroid injection group/arm since they are exposed to steroid preparation. Autologous blood injection group/arm is not exposed to any steroid preparation so total number of participants at risk is 0.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes